CLINICAL TRIAL: NCT06558045
Title: Bioequivalence Study of Rivaroxaban 20 mg Film-Coated Tablet Produced by PT Dexa Medica in Comparison With the Comparator Drug (Xarelto® 20 mg Film-Coated Tablet, Manufactured by Bayer AG, Germany, Imported by PT Bayer Indonesia, Indonesia) When Administered Under Fed Condition in Healthy Subjects
Brief Title: Bioequivalence Study of Rivaroxaban 20 mg Film-coated Tablets
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dexa Medica Group (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: BE. 787/EQL/2023
Record Dates: First submitted 2024-08-14; First posted 2024-08-16 (Actual); Last update posted 2024-08-16 (Actual); Status verified 2024-08

CONDITIONS: Healthy
MeSH Terms: interventions — Rivaroxaban

STUDY DESIGN:
Intervention Model Description: This was a bioequivalence study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test Rivaroxaban 20 mg PT Dexa Medica (Experimental): Rivaroxaban 20 mg Film-coated Tablet, produced by PT Dexa Medica, Indonesia
  Interventions: Drug: Rivaroxaban 20 mg film-coated tablet
- Reference Xarelto 20 mg Bayer (Active Comparator): Xarelto® 20 mg Film-Coated Tablet, manufactured by Bayer AG, Germany, imported by PT Bayer Indonesia, Indonesia
  Interventions: Drug: Xarelto 20 mg film-coated tablet

INTERVENTIONS:
Drug: Rivaroxaban 20 mg film-coated tablet — One tablet of the test drug was given orally 30 minutes after subjects have consumed a standardized high fat meal as breakfast
  Arms: Test Rivaroxaban 20 mg PT Dexa Medica
Drug: Xarelto 20 mg film-coated tablet — One tablet of the reference drug was given orally 30 minutes after subjects have consumed a standardized high fat meal as breakfast
  Arms: Reference Xarelto 20 mg Bayer

SUMMARY:
This study was an open-label, randomized, single-dose, two-period, two-sequence, two-way crossover study under fed conditions which included 28 healthy adult male and female subjects. The objective of this study was to compare whether the bioavailability of PT Dexa Medica's formulation of rivaroxaban 20 mg film-coated tablet is equivalent to that of the comparator drug (Xarelto® 20 mg Film-Coated Tablet, manufactured by Bayer AG, Germany, imported by PT Bayer Indonesia, Indonesia) when administered under fed condition in healthy subjects.

DETAILED DESCRIPTION:
The objective of this study was to compare whether the bioavailability of PT Dexa Medica's formulation of rivaroxaban 20 mg film-coated tablet is equivalent to that of the comparator drug (Xarelto® 20 mg Film-Coated Tablet, manufactured by Bayer AG, Germany, imported by PT Bayer Indonesia, Indonesia) when administered under fed condition in healthy subjects. This was an open-label, randomized, single-dose, two-period, two-sequence, two-way crossover study under fed conditions which included 28 healthy adult male and female subjects. The participating subjects were given orally the test drug (rivaroxaban 20 mg film-coated tablet produced by PT Dexa Medica) or the comparator drug (Xarelto® 20 mg Film-Coated Tablet, manufactured by Bayer AG, Germany, imported by PT Bayer Indonesia, Indonesia) with total 200 mL of water 30 minutes after the subjects have consumed a standardized high fat meal as breakfast meal in the first day of each period. Subjects had to ingest meal within 30 minutes or less.

Start and end of breakfast were documented. The subject's oral cavity was checked thoroughly to confirm complete medication and fluid consumption after dosing. Blood samples were drawn before taking the drug (control), and at 0.50, 1.00, 1.33, 1.67, 2.00, 2.33, 2.67, 3.00, 3.33, 3.67, 4.00, 4.33, 4.67, 5.00, 5.50, 6.00, 8.00, 12.00, 24.00 and 36.00 hours after drug administration. These blood samples were used to investigate the pharmacokinetic parameters of rivaroxaban following single dose administration. The plasma concentrations of rivaroxaban were determined by using a validated ultra-performance liquid chromatography with tandem mass spectrometry detection (UPLC-MS/MS).

ELIGIBILITY:
Inclusion Criteria:

1. Able to participate, communicate well with the investigators and willing to provide written informed consent to participate in the study.
2. Healthy male and female subjects with absence of significant disease or clinically significant abnormal laboratory values on laboratory evaluation, medical history or physical examination during screening and could be considered healthy based on the evaluation.
3. Aged 18 - 55 years inclusive.
4. Non-smokers.
5. Body mass index within 18 to 25 kg/m2.
6. Vital signs (after 10 minutes rest) must be within the following ranges:

   * Systolic blood pressure: 100 - 129 mmHg
   * Diastolic blood pressure: 60 - 84 mmHg
   * Pulse rate: 60 - 90 bpm.
7. Willing to practice abstention or contraception during the study.
8. Prothrombin time (PT) and activated partial thromboplastin time (aPTT) values should be within normal range.
9. Normal renal function with acceptable creatinine clearance (CrCl) >50 mL/min.

Exclusion Criteria:

1. History of allergy or hypersensitivity or contraindication to rivaroxaban or factor Xa inhibitors or allied drugs.
2. Pregnant or lactating female (urinary pregnancy test was applied to female subjects at screening and before taking the study drug).
3. Any major illness in the past 90 days or clinically significant ongoing chronic medical illness.
4. Presence of any clinically significant abnormal values during screening e.g. significant abnormality of liver function test (AST, ALT, alkaline phosphatase, total bilirubin, direct bilirubin ≥ 1.5 ULN), renal function test (serum creatinine concentration > 1.4 mg/dL and ureum ≥ 1.5 ULN), etc.
5. Patient with significant liver disease (severe hepatic impairment/Child Pugh C).
6. Positive Hepatitis B surface antigen (HBsAg), anti-HCV, or anti-HIV.
7. Positive result for COVID-19 rapid antigen test (this criteria only applied if the study conduct during pandemic condition).
8. Clinically significant hematology abnormalities.
9. Clinically significant electrocardiogram (ECG) abnormalities.
10. Any surgical or medical condition (present or history) which might significantly alter the absorption, distribution, metabolism or excretion of the study drug, e.g. gastrointestinal disease including gastric or duodenal ulcers or history of gastric surgery.
11. Past history of anaphylaxis or angioedema.
12. History of drug or alcohol abuse within 12 months prior to screening for this study.
13. Participation in any clinical trial within the past 90 days calculated from the last visit until this study's first dosing day.
14. History of any bleeding or coagulative disorders.
15. History of significant head or spinal cord injury or recent surgery on the brain, spinal cord or eyes.
16. Presence of difficulty in accessibility of veins in left or right arm.
17. A donation or significant blood loss within 90 days before this study's first dosing day.
18. Intake of any prescription, non-prescription drug (including hormonal contraception), food supplements or herbal medicines within 21 days of this study's first dosing day.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2023-07-06 (Actual); Primary Completion 2023-07-18 (Actual); Study Completion 2023-10-02 (Actual)

PRIMARY OUTCOMES:
AUC(0-t) | 36 hours
  Area under the plasma concentration-time curve to the last observer quantifiable concentration at time t
Cmax | 36 hours
  Maximum plasma concentration

SECONDARY OUTCOMES:
AUC(0-inf) | 36 hours
  Area under the plasma concentration-time curve extrapolated to infinitive time
T1/2 | 36 hours
  Plasma half-life
Tmax | 36 hours
  Time taken to reach maximum observed plasma concentration

CONTACTS AND LOCATIONS:
Locations (1):
- PT Equilab International, Jakarta, Indonesia